CLINICAL TRIAL: NCT05699356
Title: Surgical and Non Surgical Treatment Option in Poly Cystic Ovary Cases, A Meta Analysis Study
Brief Title: Surgical and Non Surgical Treatment Option in Poly Cystic Ovary Cases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hawala Saleh Mohammed, Resident, Sohag University
Other Study IDs: Soh-Med-22-10-03
Record Dates: First submitted 2022-10-18; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Poly Cystic Ovary Treatment for Infertility
MeSH Terms: interventions — Neoadjuvant Therapy; Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Surgical treatment of Poly cystic ovary for infertility by laparoscopic drilling: laparoscopic drilling response in Poly Cystic Ovary case
  Interventions: Procedure: laparoscopic drilling
- Non-surgical treatment of Poly cystic ovary for infertility: induction,Anti estrogen,Insulin sensitizing agent, Aromatase Inhibitor,Gonadotropin
  Interventions: Other: Non Surgical treatment
- Treatment of Poly cystic ovary for infertility by Life style modification: Life style modification response in Poly Cystic Ovary case for treatment of infertility
  Interventions: Behavioral: Treatment of Poly cystic ovary for infertility by Life style modification
- Treatment of Poly cystic ovary for infertility by Assisted reproductive technique: Assisted reproductive technique response in Poly Cystic Ovary case for treatment of infertility
  Interventions: Procedure: Treatment of Poly cystic ovary for infertility by Assisted reproductive technique
- Treatment of Poly cystic ovary for infertility by controlling menstrual disorders: Controlling menstrual disorders response in Poly Cystic Ovary case for treatment of infertility
  Interventions: Other: Non Surgical treatment
- Treatment of Poly cystic ovary for infertility by Cutaneous manifestation: Cutaneous manifestation response in Poly Cystic Ovary case for treatment of infertility
  Interventions: Other: Non Surgical treatment

INTERVENTIONS:
Other: Non Surgical treatment — Non Surgical
  Other Names: Induction, Aromatase inhibitor,Insulin sensitizing agent,Gonadotropin,Anti estrogen
  Groups: Non-surgical treatment of Poly cystic ovary for infertility; Treatment of Poly cystic ovary for infertility by Cutaneous manifestation; Treatment of Poly cystic ovary for infertility by controlling menstrual disorders
Procedure: laparoscopic drilling — Surgical intervension
  Groups: Surgical treatment of Poly cystic ovary for infertility by laparoscopic drilling
Behavioral: Treatment of Poly cystic ovary for infertility by Life style modification — Non Surgical
  Other Names: Non surgical treatment option
  Groups: Treatment of Poly cystic ovary for infertility by Life style modification
Procedure: Treatment of Poly cystic ovary for infertility by Assisted reproductive technique — Surgical intervention
  Other Names: Surgical treatment option
  Groups: Treatment of Poly cystic ovary for infertility by Assisted reproductive technique

SUMMARY:
The study will focus on treatment of Poly Cystic Ovary Syndrome patients with infertility The aim is to to find the best treatment by comparison of surgical and non surgical intervention

DETAILED DESCRIPTION:
INTRODUCTION Infertility is the failure of couples to conceive after one year of having regular unprotected coitus 1, 2&3 Globally there are 48 -186 million people cases reported with infertility. The common causes of infertility are being male factor, tubal peritoneal factor, cervical mucus, an ovulatory disorders and others causes including anti-sperm antibodies, luteal phase deficiency, diabetic mellitus, genital tract infection 1,2&4 Infertility is often multifactorial so during treatment multiple investigations should be conducted 2 Anovulation cover 30% of all infertility cases, is a complex process by which there is a failure of ovary to release mature ovarian follicles and involves a lot of potential causes 2&5 The clinical symptoms of anovulating cycles are irregular periods, light or heavy menses, deficiency of cervical mucus, Irregular Basal Body Temperature (BBT) 2&5 The common causes of anovulatory cycle is Polycystic Ovarian Syndrome (PCOS), other causes are due to hypothalamus or pituitary gland dysfunction, Premature ovarian failure, high serum estradiol in follicular phase, age above 45, hyper prolactinemia, subclinical hypothyroidism, drugs, luteinized unruptured follicles, Diabetes mellitus, athletic activity and people who do not eat and become very slim 1,2&5 Polycystic Ovarian Syndrome (PCOS) is a condition in a female of child bearing age characterized by menstrual disorders, hyperandrogenism, multiple ovarian cysts and anovulatory cycle 6 The causes of this condition are idiopathic, but the following reasons are highly suggested to be associated with PCO 6&7 Insulin resistance develop from excess insulin lead the body to produce more androgen and causing anovulatory cycle 6 women with PCOS have low grade inflammation that stimulates Poly cystic ovaries to produce androgen which can lead changes in blood vessels and heart 6 PCOS also may be due familiar susceptibility 6 The sign and symptoms of PCO are Menstrual disorders including missed period more than 35 days, infrequent period less 9 menses in a year, irregular menses light or heavy period 6&7 Hyperandrogenism manifestation like hirsutism, clitoromegaly, masculinization, severe acne, in severe form of PCO (hyperthecosis) there is deepening of voice 6, 7&8 History of infertility due to intermittently ovulation, the condition also is associate with higher chance of miscarriage 8 Polycystic ovaries presence of numerous small cysts filled with fluid in the ovaries 6&7 Majority of PCO patients are obese which worsen the symptoms of PCO 6&8 About 10 % of PCO cases have type 2 Diabetic Mellitus and 30-40 % at age of 40 have impaired glucose tolerance test 8 Sleep apnea which predispose PCO affected patients to cardiovascular disease 8 COMPLICATION OF PCO Infertility, gestational diabetes, Pregnancy induce hypertension, abortion or pre term birth, steatohepatitis, cardiovascular disease, Type 2 diabetes or prediabetes, lack of sleep, depression, thinning of hair, anxiety and eating disorder, abnormal uterine bleeding, acanthosis nigricans, armpit and under breasts, endometrial cancer a1 a2 The treatment of PCO is widely including life style modification, drug treatment, FDA safety alerts, metabolic derangements, anovulation, hirsutism, diet and activity, surgical intervention a3

ELIGIBILITY:
Inclusion Criteria:

* Infertility cases with Poly Cystic Ovary sundrome

Exclusion Criteria:

* Infertility cases not related with Poly cystic ovary

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — females on child bearing age
Study Population: Women in a child bearing age with poly cystic ovarian syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-03-28 (Estimated)

PRIMARY OUTCOMES:
The rate of ovulation after life modification | 6 months
  The study will focus on different methods of health modification like health eating, exercise and weight loss and their ability to keep hormones in normal ranges and cause ovulation
Rate of ovulation by medical treatment like Clomifene Citrate and Letrozole | 6 months
  The study also will focus on different medical treatment method like Clomifene Citrate, lentrozole for induction in ovulation
Rate of regular ovulation after laparoscopic Ovarian drilling (Surgical treatment) | 6 months
  The surgery is done to remove part of ovary through laparoscopy which results ovary to restore normal ovulation

CONTACTS AND LOCATIONS:
Locations (1):
- Suhag University hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://go.drugbank.com/drugs/DB00882